CLINICAL TRIAL: NCT01646307
Title: Effect of Atorvastatin Versus Rosuvastatin Intensive Statin Regimens on Chinese Elderly Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Effect of Atorvastatin Versus Rosuvastatin Intensive Statin Regimens on Chinese Elderly Patients Undergoing PCI
Acronym: ARISE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Vice President of Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARISE-001
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Focus of Study
MeSH Terms: interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard care group (Placebo Comparator): patients receive atorvastatin 20 mg/d
  Interventions: Drug: Atorvastatin
- intensive rosuvastatin (Active Comparator): administrated with rosuvastatin 20mg 12h prior PCI, then 10mg 2h prior PCI; followed by 10 mg/d for 30 days after PCI
  Interventions: Drug: Rosuvastatin
- intensive atorvastatin (Active Comparator): patients will be administrated with atorvastatin 80mg 12h prior PCI, then 40mg 2h prior PCI, followed by 40 mg/d for 30 days after PCI;
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin
  Arms: intensive atorvastatin; standard care group
Drug: Rosuvastatin
  Arms: intensive rosuvastatin

SUMMARY:
This randomized, open label, parallel-group study is designed to investigate whether periprocedural intensive statin therapy with atorvastatin versus rosuvastatin administration before PCI and 30-day continuous intensive treatment is superior to usual care, in terms of cardiovascular events for Chinese elderly patients.

DETAILED DESCRIPTION:
1800 elderly patients (>65 yr) with coronary artery disease undergoing elective PCI were randomized in 2:1 fashion into either intensive statin group or standard care group. Patients in intensive statin group is further randomized into two subgroups: administrated with either atorvastatin 80mg 12h prior PCI, then 40mg 2h prior PCI, followed by 40 mg/d for 30 days after PCI; or rosuvastatin 20mg 12h prior PCI, then 10mg 2h prior PCI; followed by 10 mg/d for 30 days after PCI, while the standard care group receives atorvastatin 20 mg/d. After angiography, patients who are not undergoing PCI procedure will be excluded from the study as selection failure. The last visit will be at 6 months after PCI. Clinical data such as troponin, CK-MB, Scr, CCR, ALT, AST before and 24h to 48h after procedure will be recorded. 1000 eligible patients will be finally enrolled.The study will be conducted at 12 centers in China.

ELIGIBILITY:
Inclusion Criteria:

65-80 years old Patients undergoing for elective percutaneous coronary intervention Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Patients undergoing emergency percutaneous coronary intervention
* Taking or, needing to take atorvastatin over than 20mg/d or any other equivalent statin (such as simvastatin 20mg/d, pruvastatin 40mg/d, fluvastatin 80mg/d or rovastatin 5mg/d ) in the next 6 months, or needing to take fibrates or niacins simultaneously according to investigators' judgment.
* LDL-C < 1.8mmol/L in patients without statin therapy
* Endstage congestive heart failure, or LVEF < 30%
* Active hepatic disease or hepatic dysfunction, or AST/ALT > 1.5UNL
* Myopathy or increased creatine kinase (CK>2 UNL)
* WBC < 4×109/L or PLT < 100×109/L
* Severe renal dysfunction(Scr > 3 mg/dl or 264μmol/L)
* Allergic or experienced serious adverse reaction to HMG-CoA reductase, or ineligible to take statin as investigator's judgment
* Severe aortic valve stenosis or severe mitral stenosis, Obstructive hypertrophic cardiomyopathy, pericardial diseases
* Accompanied with malignant disease or other disease, which cause life expectancy < 6 months
* Participating in other interventional clinical trials using drugs or devices
* Patients with any condition which, in the investigator's judgment, might increase the risk to the subject for any adverse event or abnormal laboratory finding

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
30-day MACCEs after PCI | 30-day after PCI
  30-day major adverse cardio- and cerebralvascular events (combined endpoints of cardiac death, myocardial infarction, stroke, stent thrombosis and target vessel revascularization ) after PCI

SECONDARY OUTCOMES:
changes in myocardial biomarkers (troponin I, Creatine kinase-MB) | 24 hours after PCI
  changes in myocardial biomarkers (troponin I, Creatine kinase-MB)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jie Zhou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China